CLINICAL TRIAL: NCT01023633
Title: A Randomized Study Of Continuous FOLFOX4 vs. FOLFOX4 in a Stop-and-Go Fashion in 1st Line Advanced Colorectal Cancer
Brief Title: OPTIMOX1 in Chinese mCRC Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Nanjing Medical University., Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Oxali04882
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Colorectal Cancer
Keywords: to investigate the efficacy and feasibility of this novel treatment strategy in Chinese mCRC patients; Primary Endpoint:DDC; Secondary Endpoint:OS, RR,DCR, PFS,safety
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: FOLFOX 4 continuous (Oxaliplatin, LV, 5-FU) (Active Comparator): The arm A (FOLFOX4 continuous arm):receive FOLFOX4 every 2 weeks until progression or for maximum 24 cycles.
  Interventions: Drug: Oxaliplatin, LV, 5-FU
- Arm B: FOLFOX4 Stop and go (Oxaliplatin, LV, 5-FU) (Experimental): The arm B will receive FOLFOX4 for 6 cycles, maintenance with 5FU/LV for 12 cycles, and reintroduction of FOLFOX4 for 6 cycles
  Interventions: Drug: Oxaliplatin, LV, 5-FU

INTERVENTIONS:
Drug: Oxaliplatin, LV, 5-FU — Arm B(Intervention arm) will receive FOLFOX4 for 6 cycles, maintenance with 5FU/LV for 12 cycles, and reintroduction of FOLFOX4 for 6 cycles.
  FOLFOX4 regimen:
  OXA 85mg/m2 , 2 hour infusion, d1 , Leucovorin 200 mg/m2 plus 5-FU 400mg IV bolus, then continuous 22 hour 600 mg/m2 infusion on day 1 and 2 Q2W
  Other Names: Eloxatin

SUMMARY:
Previous OPTIMOX1 study investigated the use of oxaliplatin discontinuation and reintroduction in a novel stop-and-go strategy. Previously untreated patients were randomly assigned to either FOLFOX4 administered every 2 weeks until progression (arm A) or FOLFOX7 for 6 cycles, maintenance without oxaliplatin for 12 cycles, and reintroduction of FOLFOX7 for another 6 cycles (arm B). Data showed that there was no significant difference in median progression-free survival (PFS) and overall survival (OS) between two arms. Furthermore, this study showed lower Grade 3 neurotoxicity rate in arm B (17.9% vs 13.3%, P = 0.12).In order to investigate the efficacy and feasibility of the novel "Stop and go" strategy in Chinese mCRC patients, Prof. Shu Yongqian in JiangShu Province Hospital plans to conduct a randomized controlled study to compare continuous FOLFOX4 vs. FOLFOX4 in a Stop-and-Go Fashion in 1st Line mCRC patients. To avoid the high oxaliplatin dosage related neurotoxicity, FOLFOX4 regimen is chosen in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed adenocarcinoma of the colon or rectum
* Unresectable metastases
* At least one bidimensionally measurable lesion of ≥ 1 cm
* No previous chemotherapy for metastatic disease; Completed at least more than 1 year oxaliplatin therapy for adjuvant treatment
* 18-75 years old
* ECOG 0-2
* Life expectancy greater than 3 months
* Hemogram: WBC≥4.0 X109/L, ANC ≥2 X109/L, PLT ≥100 X109/L, Hb ≥90g/L,
* Adequate Renal Function
* Adequate Liver Function
* Signed informed consent before the treatment

Exclusion Criteria:

* Patients with previous oxaliplatin based adjuvant chemotherapy within 1 Year
* Completely or partially bowel obstruction
* Presence of peripheral neuropathy (CTC>grade I)
* Severe mental disorder
* CNS metastasis
* With other severe disease: uncontrolled active infectious disease, uncontrolled hypertension, heart infarction within 1 year, uncontrolled high-risk arrhythmia, unstable angina
* With other malignant disease previously or concurrently
* Receive other anti-tumor treatment
* Pregnant or lactating women, or women of child bearing potential without contraceptive method.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-10; Primary Completion 2014-01 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
DDC: Duration of Disease Control | Oct2012

SECONDARY OUTCOMES:
OS, RR, PFS, DCR, safety, | Oct 2015

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The 1st Affiliated Hospital Of NanJing Medical University, Nanjing, Jiangsu
  - Zhejiang University affiliated sir run run shaw hospital, Hangzhou, Zhejiang

REFERENCES:
- [Result] Tournigand C, Cervantes A, Figer A, Lledo G, Flesch M, Buyse M, Mineur L, Carola E, Etienne PL, Rivera F, Chirivella I, Perez-Staub N, Louvet C, Andre T, Tabah-Fisch I, de Gramont A. OPTIMOX1: a randomized study of FOLFOX4 or FOLFOX7 with oxaliplatin in a stop-and-Go fashion in advanced colorectal cancer--a GERCOR study. J Clin Oncol. 2006 Jan 20;24(3):394-400. doi: 10.1200/JCO.2005.03.0106. PMID 16421419